CLINICAL TRIAL: NCT03415022
Title: A Novel Computer-Based Treatment for Social Anxiety: Target Engagement
Brief Title: Computer-Based Treatment for Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Franklin Schneier, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #7598
Record Dates: First submitted 2018-01-22; First posted 2018-01-30 (Actual); Results first posted 2020-08-11 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Social Anxiety Disorder
Keywords: SAD; Social Anxiety; Social Phobia
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Intervention Model Description: Computer-based task involving free viewing of faces and listening to music
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will not be informed as to whether a participant is randomized to 4 or 8 weeks of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4-week computer-based treatment (Experimental): A 4-week (8-sessions) course of computer-based treatment. Participants will receive treatment twice a week for four weeks.
  Interventions: Behavioral: computer-based treatment
- 8-week computer-based treatment (Experimental): An 8-week (12-sessions) course of computer-based treatment. Participants will receive treatment twice a week for four weeks, and then once a week for the subsequent four weeks.
  Interventions: Behavioral: computer-based treatment

INTERVENTIONS:
Behavioral: computer-based treatment — 30 minute sessions of free viewing of faces and listening to music

SUMMARY:
The present study is an open trial that seeks to examine the feasibility, acceptability, mechanism, and efficacy of a recently developed computer-based therapy in individuals with social anxiety disorder (SAD)

DETAILED DESCRIPTION:
This randomized clinical trial examines the feasibility, acceptability, mechanism, and relative efficacy of two "doses" (standard 4-week/8 session vs. extended 8-week/12-session) of a recently developed computer-based therapy in individuals with social anxiety disorder (SAD). The purpose of this study is to assess whether a brief computer-based research treatment, provided in 30 minutes sessions, helps improve social anxiety symptoms, and by what mechanism. The study will also assess the effect of research treatments on brain activity using magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 and 60
* Current primary diagnosis of SAD
* Score of at least 50 on the Liebowitz Social Anxiety Scale (Self-rated version)
* Fluent in English and willing and able to give informed written consent and participate responsibly in the protocol
* Normal or corrected-to-normal vision

Exclusion Criteria:

* Present or past psychotic episode, psychotic disorder, schizophrenia, schizoaffective disorder, or bipolar disorder
* Current severe depression
* Suicidal ideation or behavior
* Current diagnosis of posttraumatic stress disorder, obsessive-compulsive disorder, bipolar disorder, manic episode or tic disorder
* Current or past organic mental disorder, seizure disorder, epilepsy or brain injury
* Current unstable or untreated medical illness
* Severe alcohol use disorder, severe cannabis use disorder, and any severity of other substance use disorder (except nicotine use disorders allowed)
* Use of psychiatric medication in the past month other than a stable dose of selective serotonin reuptake inhibitors (SSRIs) for a least 3 months
* Any concurrent cognitive behavioral therapy; other psychotherapy that was initiated in the past 3 months
* Pregnancy, or plans to become pregnant during the period of the study - will be assessed by urine
* Contraindication to MRI scanning:
* Paramagnetic metallic implants or devices contraindicating magnetic resonance imaging or any other non-removable paramagnetic metal in the body (e.g. pacemaker, paramagnetic metallic prosthesis, surgical clips, shrapnel, necessity for constant medicinal patch, some tattoos)
* Being unable to tolerate the scanning procedures (i.e., severe obesity, claustrophobia)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Schneier, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the National Database for Clinical Trials related to Mental Illness (NDCT). We will generate a Global Unique Identifier (GUID) for each participant. The key clinical rating scale measures (LSAS, SPIN, QLESQ, HRSD) are all included.
Supporting Information: Analytic Code
Time Frame: Raw data will be submitted semi-annually every January 15 and July 15.
Access Criteria: see URL below for criteria
URL: https://nda.nih.gov/

REFERENCES:
- [Background] Chevallier C, Tonge N, Safra L, Kahn D, Kohls G, Miller J, Schultz RT. Measuring Social Motivation Using Signal Detection and Reward Responsiveness. PLoS One. 2016 Dec 1;11(12):e0167024. doi: 10.1371/journal.pone.0167024. eCollection 2016. PMID 27907025
- [Background] Cisler JM, Koster EH. Mechanisms of attentional biases towards threat in anxiety disorders: An integrative review. Clin Psychol Rev. 2010 Mar;30(2):203-16. doi: 10.1016/j.cpr.2009.11.003. Epub 2009 Dec 14. PMID 20005616
- [Background] Gur RC, Schroeder L, Turner T, McGrath C, Chan RM, Turetsky BI, Alsop D, Maldjian J, Gur RE. Brain activation during facial emotion processing. Neuroimage. 2002 Jul;16(3 Pt 1):651-62. doi: 10.1006/nimg.2002.1097. PMID 12169250
- [Background] Heeren A, Mogoase C, Philippot P, McNally RJ. Attention bias modification for social anxiety: A systematic review and meta-analysis. Clin Psychol Rev. 2015 Aug;40:76-90. doi: 10.1016/j.cpr.2015.06.001. Epub 2015 Jun 6. PMID 26080314
- [Background] Klumpp H, Angstadt M, Phan KL. Shifting the focus of attention modulates amygdala and anterior cingulate cortex reactivity to emotional faces. Neurosci Lett. 2012 Apr 18;514(2):210-3. doi: 10.1016/j.neulet.2012.03.003. Epub 2012 Mar 8. PMID 22425719
- [Background] Klumpp H, Post D, Angstadt M, Fitzgerald DA, Phan KL. Anterior cingulate cortex and insula response during indirect and direct processing of emotional faces in generalized social anxiety disorder. Biol Mood Anxiety Disord. 2013 Apr 2;3:7. doi: 10.1186/2045-5380-3-7. eCollection 2013. PMID 23547713
- [Background] Lazarov A, Abend R, Bar-Haim Y. Social anxiety is related to increased dwell time on socially threatening faces. J Affect Disord. 2016 Mar 15;193:282-8. doi: 10.1016/j.jad.2016.01.007. Epub 2016 Jan 12. PMID 26774515
- [Background] Lazarov A, Pine DS, Bar-Haim Y. Gaze-Contingent Music Reward Therapy for Social Anxiety Disorder: A Randomized Controlled Trial. Am J Psychiatry. 2017 Jul 1;174(7):649-656. doi: 10.1176/appi.ajp.2016.16080894. Epub 2017 Jan 20. PMID 28103714
- [Background] Linetzky M, Pergamin-Hight L, Pine DS, Bar-Haim Y. Quantitative evaluation of the clinical efficacy of attention bias modification treatment for anxiety disorders. Depress Anxiety. 2015 Jun;32(6):383-91. doi: 10.1002/da.22344. Epub 2015 Feb 24. PMID 25708991
- [Background] Mogoase C, David D, Koster EH. Clinical efficacy of attentional bias modification procedures: an updated meta-analysis. J Clin Psychol. 2014 Dec;70(12):1133-57. doi: 10.1002/jclp.22081. Epub 2014 Mar 20. PMID 24652823
- [Background] Morrison AS, Heimberg RG. Social anxiety and social anxiety disorder. Annu Rev Clin Psychol. 2013;9:249-74. doi: 10.1146/annurev-clinpsy-050212-185631. PMID 23537485
- [Background] Richey JA, Rittenberg A, Hughes L, Damiano CR, Sabatino A, Miller S, Hanna E, Bodfish JW, Dichter GS. Common and distinct neural features of social and non-social reward processing in autism and social anxiety disorder. Soc Cogn Affect Neurosci. 2014 Mar;9(3):367-77. doi: 10.1093/scan/nss146. Epub 2012 Dec 7. PMID 23223206
- [Background] Spreckelmeyer KN, Krach S, Kohls G, Rademacher L, Irmak A, Konrad K, Kircher T, Grunder G. Anticipation of monetary and social reward differently activates mesolimbic brain structures in men and women. Soc Cogn Affect Neurosci. 2009 Jun;4(2):158-65. doi: 10.1093/scan/nsn051. Epub 2009 Jan 27. PMID 19174537
- [Background] Van Bockstaele B, Verschuere B, Tibboel H, De Houwer J, Crombez G, Koster EH. A review of current evidence for the causal impact of attentional bias on fear and anxiety. Psychol Bull. 2014 May;140(3):682-721. doi: 10.1037/a0034834. Epub 2013 Nov 4. PMID 24188418

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 participants discontinued the study after initial evaluation but before treatment randomization:
  * 5 discontinued due to scheduling difficulties
  * 2 discontinued due to COVID-19 research suspension
  * 2 discontinued due to difficulties calibrating eye tracker used for treatment sessions
Period: Overall Study
Arm/Group | 4-week Computer-based Treatment | 8-week Computer-based Treatment
Started | 21 | 20
Completed | 16 | 15
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — COVID-19 Suspension | 2 | 3
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants who started treatment sessions
Groups:
- Total: Total of all reporting groups
Arm/Group | 4-week Computer-based Treatment | 8-week Computer-based Treatment | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (5.08) | 29.15 (7.13) | 28.61 (6.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 10 | 6 | 16
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41
Liebowitz Social Anxiety Scale [Mean (Standard Deviation); unit: units on a scale] — This clinician-reported scale is used to assess social anxiety. Participants were provided with a list of 24 social situations and rated their anxiety in that situation on a scale from 0-3, and their avoidance of that situation on a scale from 0-3. The measure is scored by adding the total of anxiety ratings and avoidance ratings (scores range from 0-144).
  units on a scale | 83.8 (16.81) | 87.6 (11.32) | 86.05 (14.28)

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Dwell Time on Threat Faces
Description: Percent dwell time on threat faces was computed as the ratio of gaze dwell time on threat faces to total dwell time on all faces as measured by eye tracking during treatment sessions. Change in percent dwell time is the value at week 8 minus value at baseline.
Time Frame: baseline to week 8
Measure: Mean (Standard Deviation); unit: percentage of dwell time on threat faces
Arm/Group | 4-week Computer-based Treatment | 8-week Computer-based Treatment
Number analyzed (Participants) | 16 | 15
percentage of dwell time on threat faces | 20.7 (20.6) | 27.1 (17.6)

2. Primary Outcome: Change in Total Score of Liebowitz Social Anxiety Scale (LSAS)
Description: Clinician-rated scale scoring anxiety (0, none to 3, severe) and avoidance (0,none to 3, severe) in 24 social situations for a total score of 0 to 144. Higher scores indicate greater social anxiety.
Time Frame: Baseline to week 8
Population: Participants who completed 8 weeks of study participation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-week Computer-based Treatment | 8-week Computer-based Treatment
Number analyzed (Participants) | 16 | 15
score on a scale | 23.68 (32.44) | 22.38 (22.87)

3. Secondary Outcome: Change in Total Score of Social Phobia Inventory (SPIN)
Description: The Social Phobia Inventory (SPIN) is a self-rated questionnaire used to assess severity of social anxiety disorder. 17 items related to social anxiety each rated on a score of 0 to 4, with a minimum total score of 0 (least social anxiety), and a maximum total score of 68 (most social anxiety).
Time Frame: baseline to week 8
Population: participants with 8 weeks of assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-week Computer-based Treatment | 8-week Computer-based Treatment
Number analyzed (Participants) | 16 | 15
score on a scale | 17.7 (18.5) | 10.1 (13.5)

4. Secondary Outcome: Change in Total Score of Quality of Life Enjoyment & Satisfaction Questionnaire
Description: Quality of Life Enjoyment & Satisfaction Questionnaire (Q-LES-Q): self-rated assessment of quality of life. 16 items related to life quality, each rated on a score of 1 (very poor) to 5 (very good), with a minimum total score of 16, and a maximum total score of 80.
Time Frame: baseline to week 8
Population: participants who completed 8 weeks of assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 4-week Computer-based Treatment | 8-week Computer-based Treatment
Number analyzed (Participants) | 16 | 15
score on a scale | -8.8 (15.3) | -4.8 (12.4)

5. Secondary Outcome: Change in Total Score of the Revised Social Anhedonia Scale
Description: 40-item self-rated social anhedonia scale. Items are comprised of statements that participants agree or disagree with, by answering "yes"(1), or "no"(0), with some items reverse-coded. The minimum score is 0 (least social anhedonia); maximum score is 40 (most social anhedonia)
Time Frame: baseline to week 8
Population: participants who completed 8 weeks of assessments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 4-week Computer-based Treatment | 8-week Computer-based Treatment
Number analyzed (Participants) | 16 | 15
units on a scale | 1.7 (5.6) | 1.8 (4.9)

6. Secondary Outcome: Change in Total Score of the Snaith Hamilton Pleasure Scale
Description: Snaith Hamilton Pleasure Scale (SHAPS). Fourteen-item self-rated anhedonia scale. Items are comprised of statements that participants rate as "strongly disagree" (1), "disagree" (2), "agree" (3), or "strongly agree" (4). The lowest possible score was 14, the highest possible score was 56 (greatest anhedonia)
Time Frame: baseline to week 8
Population: participants who completed 8 weeks of assessments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 4-week Computer-based Treatment | 8-week Computer-based Treatment
Number analyzed (Participants) | 16 | 15
units on a scale | 2.2 (6.2) | -1.0 (5.8)

7. Secondary Outcome: Change in Total Score of the Hamilton Rating Scale for Depression - 17 Item Version
Description: Hamilton Rating Scale for Depression -17 item version. This standard scale will be used to assess severity of depression, minimum score is 0 (least depression); maximum score is 50 (greatest depression).
Time Frame: baseline to week 8
Population: participants who completed 8 weeks of assessments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 4-week Computer-based Treatment | 8-week Computer-based Treatment
Number analyzed (Participants) | 16 | 15
units on a scale | 1.8 (4.4) | 1.8 (5.8)

8. Secondary Outcome: Clinical Global Impression-Change Scale
Description: Clinical Global Impression-Change Scale: An observer rating of overall clinical change, with rating from 1 (very much improved) to 7 (very much worse). Responder category is defined by a score of 1 or 2.
Time Frame: week 8
Population: participants who completed 8 weeks of assessments
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 4-week Computer-based Treatment | 8-week Computer-based Treatment
Number analyzed (Participants) | 16 | 15
units on a scale | 2.8 (1.2) | 2.7 (0.9)

ADVERSE EVENTS:
Time Frame: 20 weeks (8 weeks of active treatment phase and 3 month follow-up phase)
Arm/Group | 4-week Computer-based Treatment | 8-week Computer-based Treatment
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT03415022/Prot_SAP_000.pdf